CLINICAL TRIAL: NCT04049370
Title: Examination of the Standardized Use of the Pulmonary Embolism SOP in the Clinical Routine of the Emergency Department in Respect of the QEST Criteria (Quality, Efficacy, Safety and Transparency).
Brief Title: Examination of the Standardized Use of the Pulmonary Embolism SOP in the Clinical Routine of the Emergency Department.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Evangelos Giannitsis, Principle Investigator, Heidelberg University
Other Study IDs: SOP_PE_Giannitsis
Record Dates: First submitted 2019-07-29; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; clinical decision tool; standard operating procedure
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective data collection of the "actual state": Retrospective data collection of the "actual state" 6 months prior to August 2019.
  Interventions: Other: No intervention
- Prospective data collection: Prospective data collection after implementation of the quality assurance measure for another 6 months (SOP as clinical decision tool into the electronic database of the CPU).

INTERVENTIONS:
Other: No intervention — Assessment of the "actual state" prior to implementation of the SOP as clinical decision tool into the electronic database of the chest pain unit.
  Groups: Retrospective data collection of the "actual state"

SUMMARY:
Usage of a guideline-compliant SOP in each chest pain unit (CPU) is instrumental in establishing the diagnosis of a pulmonary embolism without time delay. With the integration of this SOP as a "clinical decision tool" (CDT) into the electronic database of the CPU, the standardized application of the pulmonary embolism SOP in the clinical routine of the CPU will be tested using a retro- and prospective approach.

DETAILED DESCRIPTION:
Summary:

The increasing number of patients in the emergency departments in recent years extends the time until diagnosis and treatment initiation and thus represents a serious problem in patient care and for the treating physician. This also includes patients with acute pulmonary embolism (PE), which is one of the most common differential diagnoses of patients presenting with unclear dyspnea, chest pain or other symptoms in the emergency department. Due to the potentially serious clinical outcome with a high overall mortality rate of > 10%, rapid diagnosis and initiation of therapy is essential.

The current guidelines of the European Society of Cardiology for the diagnosis and treatment of acute PE recommend a stringent diagnostic algorithm that includes clinical parameters as well as risk scores for estimating the pretest probability. Depending of their results the further diagnostic pathway by D-Dimer testing and / or CT angiography is chosen.

The aim of the present study is to examine the standardized application of guideline recommendations of the European Society of Cardiology (ESC). The diagnostic procedures were defined for the CPU of the University Hospital Heidelberg in a standard operating procedure (SOP). In the planned retrospective study, the implementation of this SOP will be examined on the basis of the QEST criteria (quality, efficacy, safety and transparency). Data for the "actual condition" are collected retrospectively for 6 months prior to August 2019, thereafter for another 6 months after implementation of the quality assurance measure.

Introduction and fundamental principles:

Acute pulmonary embolism (PE), with a prevalence of 1.22-1.83 persons per 100,000 population, is the third most common cardiovascular disease and represents a serious disease with a 30-day mortality from potential right ventricular dysfunction with cardiogenic shock estimated at 16%. Approximately 65% of all deaths occur within the first hours after admission. The prognosis of pulmonary embolism is highly variable and depends in particular on the severity of the hemodynamic impairment as well as on concomitant morbidities.

Due to multiple and sometimes non-specific symptoms, the diagnosis of PE poses a clinical challenge and requires much clinical experience in order not to overlook the diagnosis. Clinical scores (Well's Score, Geneva Score, modified Geneva Score) and the overall clinical impression (gestalt) are used to estimate the pretest probability. The current guidelines of the European Society of Cardiology on the diagnosis and management of acute pulmonary embolism recommend a stringent diagnostic algorithm which includes clinical parameters and the above-mentioned risk scores for the assessment of the pretest probability and on the basis of them further diagnostic steps by D-dimer measurement and / or CT angiography. With a low pretest probability, a pulmonary embolism can be excluded with a probability of nearly 100%. On the other hand, if there is a high pretest probability, no D-dimer determination should be made, as even a negative result will not be able to exclude the diagnosis with certainty. The procedure for a mean pretest probability depends on the D-dimer test used. Determination of D-dimers should only be undertaken if an analytically sensitive D-dimer test is present, which is ideally authorized for the purpose of diagnostic exclusion. The central laboratory of the University Hospital of Heidelberg uses the Siemens Liason D-Dimer test, which is considered one of the most sensitive tests. From the diagnostic procedure, a sequential pathway is recommended in which first the pre-test probability and then - depending on the estimate - the D-dimer determination follows. If pulmonary embolism cannot be ruled out, further diagnostic imaging should be provided. CT angiography with a multi-slice device (> 16-slices) is considered the diagnostic gold standard.

However, the guideline-compliant algorithm for the diagnosis of PE has so far only been investigated in a few prospective, randomized studies.

The aim of the present study is to test the standardized use of the pulmonary embolism SOP in the clinical routine of the CPU compared to the "actual state". Currently, the attending physician has unrestricted access to the determination of the D-dimer concentration, and the diagnostic process continues to be carried out at clinical discretion. These two approaches are to be tested and compared with regard to the QEST criteria (quality, efficacy, safety and transparency).

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 with suspected pulmonary embolism in the CPU (with or without D-dimer determination)

Exclusion Criteria:

* Patients in whom the determination of the D-dimer concentration was made for other reasons, such as venous thrombosis or aortic syndrome
* Patients who have been suspected to have a pulmonary embolism already before presenting in the CPU
* Patients with confirmed diagnosis or already measured D-dimers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises all patients presenting in the CPU with signs and symptoms of a pulmonary embolism (no preselection of patients).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Guideline adherence | 6 months
  • Percent guideline adherence or violation of guideline recommendations (quality)
Appropriateness of CT imaging | 6 months
  • Ratio of diagnostic CT: total CT
Missed pulmonary embolism | 6 months
  * Number of indicated but not performed CT examinations
  * Number of unnecessary CT at low pretest probability

SECONDARY OUTCOMES:
Appropriate biomarker utilization | 6 months
  • Ratio of effective D-dimers: total D-dimers at low pretest probability
Inappropriate biomarker utilization | 6 months
  • Number of unnecessary D-dimers at high pretest probability
efficacy of CT imaging | 6 months
  • Number of unnecessary CT at low pretest probability

OTHER OUTCOMES:
Length of stay in emergency department | 6 months
  • Time spent in the CPU,
Time to diagnosis | 6 months
  duration from hospital admission to CT

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giannitsis, Prof., Principal Investigator — Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided